CLINICAL TRIAL: NCT01003782
Title: Routine Bile Collection for Microbiological Analysis During Cholangiography and Its Impact on Management of Cholangitis: Results of a Prospective Study
Brief Title: Routine Bile Collection for Microbiological Analysis During Cholangiography
Acronym: ERCP
Status: Completed | Type: Observational
Sponsor: Hannover Medical School (Other)
Responsible Party: Tim Lankisch, Department of Gastroenterology, Hepatology and Endcrinology
Other Study IDs: MAERCP
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2009-10-29 (Estimated); Status verified 2009-10

CONDITIONS: Cholangitis
Keywords: cholangitis; antibiotic; bacteriobilia; bile; ERCP
MeSH Terms: conditions — Cholangitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bile samples for microbiological analysis
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Antibiotic treatment of cholangitis often remains insufficient due to inappropriate antibiotic use or bacterial resistance.

Objective: To evaluate the role of routine bile collection during endoscopic retrograde cholangiography (ERC) or percutaneous transhepatic cholangiography (PTC) for microbiological analysis in the antibiotic management of cholangitis and to identify risk factors of microbial growth.

Design: Prospective, observational, diagnostic study.

Setting: Hannover Medical School, Hannover, Germany. Patients and Interventions: Consecutive patients undergoing ERC/PTC for biliary complications after orthotopic liver transplantation , malignancy, primary sclerosing cholangitis, benign strictures and choledocholithiasis.

Main outcome measurements: Microbiological examination of bile samples

ELIGIBILITY:
Inclusion Criteria:

* age above 18 years
* written informed consent

Exclusion Criteria:

* age under 18 years
* no written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients presenting to Endoscopic retrograde cholangiography
Sampling Method: Probability Sample
Dates: Start 2008-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Hannover Medical school, Hanover, Germany